CLINICAL TRIAL: NCT05878184
Title: A Phase 1 Study Evaluating SC291, a Hypoimmune, Allogeneic CD19-directed CAR T Cell Therapy, in Relapsed and/or Refractory B-cell Malignancies (ARDENT)
Brief Title: Study Evaluating SC291 in Subjects With r/r B-cell Malignancies (ARDENT)
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Sana Biotechnology (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SC291-101
Record Dates: First submitted 2023-04-28; First posted 2023-05-26 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-09

CONDITIONS: Non Hodgkin Lymphoma; Chronic Lymphocytic Leukemia
Keywords: Large B cell lymphoma; CAR T Cell Therapy; Mantle cell lymphoma; Indolent follicular lymphoma; Marginal zone lymphoma; High-grade B cell lymphoma; Primary mediastinal B cell lymphoma; Diffuse large B cell lymphoma; Non-Hodgkin's Lymphoma; Chronic Lymphocytic Leukemia; Allogeneic; Hypoimmune; CD19
MeSH Terms: conditions — Lymphoma, Non-Hodgkin; Leukemia, Lymphocytic, Chronic, B-Cell; Lymphoma, Mantle-Cell; Lymphoma, B-Cell, Marginal Zone; Lymphoma, Large B-Cell, Diffuse | interventions — Cyclophosphamide; fludarabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- SC291 Plus Chemotherapy Regimen (Experimental): A conditioning chemotherapy regimen of fludarabine and cyclophosphamide will be administered followed by investigational treatment with SC291
  Interventions: Drug: SC291

INTERVENTIONS:
Drug: SC291 — SC291 is an allogeneic CAR-T cell therapy
  Other Names: Cyclophosphamide; Fludarabine

SUMMARY:
SC291-101 is a Phase 1 study to evaluate SC291 safety and tolerability, anti-tumor activity, cellular kinetics, immunogenicity, and exploratory biomarkers.

DETAILED DESCRIPTION:
This is an open-label, single arm, Phase 1, first-in-human (FIH) study to evaluate the safety and tolerability of SC291 administered intravenously (IV) following a standard lymphodepleting chemotherapy regimen of cyclophosphamide and fludarabine in subjects with NHL or CLL who have received two or more prior systemic treatments per standard of care (or after autologous stem cell transplant [ASCT] for NHL). This study will be conducted in 2 parts. Phase 1a: dose finding using a 3+3 design in subjects with NHL or CLL. Phase 1b: dose expansion to further evaluate safety and efficacy at the RP2D in subjects with LBCL and CLL.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects aged 18-80 years at the time of signing informed consent.
* Diagnosis of NHL (WHO 2016 criteria) or CLL (iwCLL criteria), including:
* Large B-cell lymphoma, including diffuse large B-cell lymphoma (DLBCL) not otherwise - - specified (including DLBCL arising from indolent lymphoma), primary mediastinal large -- - B-cell lymphoma, high grade B-cell lymphoma, follicular lymphoma grade 3B
* Follicular lymphoma (dose escalation only except for follicular lymphoma grade 3B)
* Marginal zone lymphoma (dose escalation only)
* Mantle cell lymphoma (dose escalation only)
* CLL or SLL
* Relapsed/refractory disease after at least 2 prior systemic regimens per standard of care or after autologous stem cell transplant
* ECOG performance status of 0 or 1.
* At least one measurable lesion per Lugano Classification (NHL); CLL subjects must meet iwCLL treatment criteria
* Life expectancy ≥12 weeks

Exclusion Criteria:

* Prior anti-CD19 therapy including CD19-directed CAR T treatment or other CD19-directed antibody or cell therapy (e.g., NK cell). (Part 2 dose expansion only - prior approved CD19-directed CAR T therapy required)
* History of primary central nervous system (CNS) lymphoma or presence of CNS metastases
* Systemic anticancer therapy (including platinum-based chemotherapies and I/O therapies) or radiotherapy within 14 days of SC291 (28 days for biologics)
* Autologous HSCT within 6 weeks of treatment with SC291 (or allogeneic HSCT at any time).
* Active autoimmune disease or any other diseases requiring immunosuppressive therapy or corticosteroid therapy (defined as >20 mg/day prednisone or equivalent).
* History or presence of cardiac or CNS disorders as defined in the protocol

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2023-05-02 (Actual); Primary Completion 2025-11-04 (Estimated); Study Completion 2038-11-04 (Estimated)

PRIMARY OUTCOMES:
Evaluate safety and tolerability of SC291 | 24 months
  Safety and Tolerability: Proportion of subjects experiencing adverse events and dose-limiting toxicities

SECONDARY OUTCOMES:
Evaluate preliminary anti-tumor activity of SC291 | 24 months
  Preliminary anti-tumor activity: Proportion of subjects with an objective response (including partial response or complete response)
Evaluate cellular kinetics and persistence of SC291 | 24 months
  Cellular kinetics-related parameters evaluated by CAR T cell copy number
Evaluate cellular kinetics and persistence of SC291 | 24 months
  Cellular kinetics related peak (Cmax) in peripheral blood
Evaluate cellular kinetics and persistence of SC291 | 24 months
  Area under the concentration time curve (AUC) in peripheral blood
Evaluate host immunogenicity to SC291 | 24 months
  Incidence of anti-CD19-directed CAR antibodies

CONTACTS AND LOCATIONS:
Overall Officials: John Gerecitano, MD, PhD, Study Director — Sana Biotechnology, Inc.
Locations (10):
- United States (7):
  - City of Hope, Duarte, California
  - Stanford Cancer Institute, Palo Alto, California
  - Northside Hospital, Atlanta, Georgia
  - University of Kansas Medical Center, Fairway, Kansas
  - Karmanos Cancer Institute, Detroit, Michigan
  - University of Nebraska Medical Center, Omaha, Nebraska
  - MD Anderson Cancer Center, Houston, Texas
- Australia (3):
  - Royal Adelaide Hospital, Adelaide, South Australia
  - Peter MacCallum Cancer Centre, Melbourne, Victoria
  - Linear Clinical Research Ltd, Nedlands, Western Australia

IPD SHARING:
Plan to Share IPD: No